CLINICAL TRIAL: NCT06101485
Title: Future Patient - Telerehabilitering af Patienter Med Atrieflimren (FP-AF)
Brief Title: Future Patient - Telerehabilitation of Patients With Atrial Fibrillation
Acronym: (FP-AF)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aalborg University (Other)
Collaborators: Department of Cardiology, Viborg Regional Hospital (Unknown); Department of Cardiology, Silkeborg Regional Hospital (Unknown); Center for Innovative Medical Technologies (CIMT), Odense University Hospital (Unknown); Laboratory for Welfare Technology, Department of Health Science and Technology, Aalborg University (Unknown)
Responsible Party: Principal Investigator, Birthe Dinesen, Professor, Aalborg University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N-20220056
Record Dates: First submitted 2023-06-26; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Atrial Fibrillation
Keywords: Telerehabilitation; Quality of life; Cardiac patients; Atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Telerehabilitation

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation group (Experimental): The telerehabilitation group (n=104) will participate in the FP-AF program for 16 weeks. The program is administered by the AF clinics and the healthcare centers (HC) in Viborg, Skive and Silkeborg Municipalities. After enrollment, the patients will have an individual meeting with the project nurse. Here the patient (and relatives, if necessary) will be instructed in the use of the technologies and an individual plan will be formulated for the AF patient's telerehabilitation. After participation in 16 weeks the patients start a 12 weeks follow-up period, where they will only measure steps and have access to the Heartportal on their own devices.
  Interventions: Device: Telerehabilitation
- Conventional rehabilitation (No Intervention): The control group (n=104) will follow the conventional care regime in the AF clinic and will not have contact to the project nurse. When the AF patients are in a stable condition, they will be followed by their general practitioner (GP). The control group will be in the study for 28 weeks.

INTERVENTIONS:
Device: Telerehabilitation — Telerehabilitation platform: Hjerteportalen, blood pressure monitor (iHealth(neo/BP5s), weight scale (iHealth Lina), Activity tracker (FitBit inspire 3), ECG monitor (AliveCor KardiaMobile), sleep sensor (Emfit QS), video consultation (VDX by MedCom)
  Arms: Telerehabilitation group

SUMMARY:
This project has focus on patients with atrial fibrillation testing a telerehabilitation program for patients with atrial fibrillation.

DETAILED DESCRIPTION:
The overall aim of the FP-AF program is to increase quality of life by giving the patients and relatives more knowledge about atrial fibrillation, its symptoms, and the issues of living with atrial fibrillation in everyday life. The specific aims are to individualize the rehabilitation process and help the patients and relatives develop their own self-management strategies using their own clinical data and their enhanced knowledge about AF.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with atrial fibrillation
* Adults over 18 years
* Living in Skive, Viborg or Silkeborg Municipalities
* Living at home and capable of caring for themselves
* Have basic computer skills or having a relative/friend with basic computer skills

Exclusion Criteria:

* Pregnancy
* Refusal or inability to cooperate; or patient not does not speak, read or understand Danish
* Life expectancy less than a year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes in AF specific health-related quality of life | For both intervention and control group: QoL will be measured at baseline, end of telerehabilitation (16 weeks) and after 28 weeks
  The Atrial Fibrillation Effect on quality of life questionnaire (AFEQT) is a 20-item self-administered questionnaire designed to assess the impact of AF on the patients' health-related quality of life (HRQoL) across symptoms, daily activities, treatment concerns, and treatment satisfaction. Scores range from 0-100, with higher scores indicating better HRQoL

SECONDARY OUTCOMES:
Changes in AF knowledge | For both intervention and control group: To be measured at baseline, end of telerehabilitation (16 weeks) and after 28 weeks
  Changes in AF knowledge assessed by the Jessa Atrial Fibrillation Knowledge Questionnaire (JAKQ). JAKQ is a 16-item scale used to assess the knowledge the patients have about their illness. For every item, false responses or "I do not know" responses is scored as 0 and the correct responses are scored as 1. The total score of the scale is calculated by adding up the scores from each item. A score between 0% and 100% will be generated. 100% is the best possible score, meaning all questions was answered correctly.
Measurement of weight | Intervention group: Weight will be measured at baseline, twice a week, and as needed up to 16 weeks
  Intervention group: Weight (Kilograms)
Measurement of bloodpressure | Intervention group: Bloodpressure will be measured at baseline, twice a week, and as needed up to 16 weeks
  Intervention group: Bloodpressure (mmHG) (systolic and diastolic)
Measurement of pulse | Intervention group: Pulse will be measured at baseline, everyday, and as needed up to 16 weeks
  Intervention group: Pulse (numbers per minute)
Measurement of steps | Intervention group: Steps will be measured from the date of randomization, everyday to end follow up (28 weeks)
  Intervention group: numbers of steps taken
Measurement of sleep | Intervention group: Sleep will be measured every day up to 16 weeks
  Intervention group: Sleep (numbers of hours per night)
Measurement of heart rhythm | Intervention group: ECG wil be measured at baseline, twice a week, and as needed up to 16 weeks
  Intervention group: Electrocardiogram (ECG)
Changes in anxiety and depression | Both intervention and control group: At baseline, end of telerehabilitation (16 weeks) and after 28 weeks.
  The patients degree of anxiety and depression measured by the Hospital Anxiety and Depression Scale (HADS). The patient will get a score between 0 and 21 for both depression and anxiety ( 0-7 points: low level of symptoms for depression or anxiety, 8-10 points: moderate level of symptoms for depression or anxiety, 11-21 points: high level of symptoms for depression or anxiety)
Changes in motivation | Both intervention and control group: At baseline, end of telerehabilitation (16 weeks) and after 28 weeks.
  Changes in motivation measured by Healthcare, Self-Determination Theory Questionnaire Packet (HC-SDTQ) comprised of Treatment Self-Regulation Questionnaire (TSRQ); Perceived Competence Scale (PCS); and Health Care Climate Questionnaire (HCCQ). TSRQ is used to assess different forms of motivation within the self determination theory (STD). The patients are asked to answer 15 questions regarding why they either follow or do not follow their treatment by marking to which degree each reason is true on a scale form 1 to 7, with 7 being very true.
Changes in motivation | Both intervention and control group: At baseline, end of telerehabilitation (16 weeks) and after 28 weeks.
  Changes in motivation measured by Healthcare, Self-Determination Theory Questionnaire Packet (HC-SDTQ) comprised of Treatment Self-Regulation Questionnaire (TSRQ); Perceived Competence Scale (PCS); and Health Care Climate Questionnaire (HCCQ). The PCS is used to assess the patients feeling of competence about engaging in, or maintaining, a healthier behavior. It is a short 4-item questionnaire where the patients have to indicate the extent to which each reason is true on a scale from 1 to 7, with 7 indicating 'very true'.
Changes in motivation | Both intervention and control group: At baseline, end of telerehabilitation (16 weeks) and after 28 weeks.
  Changes in motivation measured by Healthcare, Self-Determination Theory Questionnaire Packet (HC-SDTQ) comprised of Treatment Self-Regulation Questionnaire (TSRQ); Perceived Competence Scale (PCS); and Health Care Climate Questionnaire (HCCQ). The HCCQC is used to assess the degree to which a patient perceives their health care providers are supportive of their autonomy. It is a 6-item questionnaire where the patients have to indicate the extent to which each reason is true on a scale from 1 to 7, with 7 indicating 'very true'.
Burden of AF | Both intervention and control group: At baseline, end of telerehabilitation (16 weeks) and after 28 weeks.
  AF burden measured by the arrhythmia-specific questionnaire in Tachycardia and Arrhythmia (ASTA questionnaire). ASTA is used to assess symptoms and health-related quality of life(HRQoL) in patients with different forms of arrythmias, including AF. It is structured into three sections:Part I assesses demographic data such as the last episode of arrhythmia, current medication, and the presence of arrhythmia at the time of follow-up; Part II measures the arrhythmia-specific symptom burden; and part III assesses HRQoL. The ASTA 9-item symptom scale and the 13-item HRQoL scale utilize a four-point Likert-type scale, ranging from 'No' to 'Yes, a lot.' The total score ranges from 0 to 100, with a higher score indicating a greater symptom burden or a more negative impact on HRQoL.
Patients' and relatives' expectations for and experiences with participation in the tele-rehabilitation program (including the Heartportal) | Intervention group: Interviews at end of telerehabilitation (16 weeks) and logfiles and observation at end follow up (28 weeks)
  Perspectives and experiences of patients and relatives participating in the FP-AF program (including the Heartportal) measured by interviews with patients and relatives.
Patients' and relatives' expectations for and experiences with participation in the tele-rehabilitation program (including the Heartportal) | Intervention group: Interviews at end of telerehabilitation (16 weeks) and logfiles and observation at end follow up (28 weeks)
  Patients and relatives use of HeartPortal measured in logfiles on use & via observation in everyday life
Healthcare professionals' experiences with workflows and collaboration with each other in the telerehabilitation program. | Intervention group: End of telerehabilitation (16 weeks)
  Perspectives and experiences of healthcare professionals participating in the FP-AF program through interviews.
Healthcare professionals' experiences with workflows and collaboration with each other in the telerehabilitation program. | Intervention group: End of telerehabilitation (16 weeks)
  Perspectives and experiences of healthcare professionals participating in the FP-AF program by observation of use of Heartportal
Cost-effectiveness analysis of the FP-AF telerehabilitation program compared to conventional care | Both intervention and control group: at the end of telerehabilitation (16 weeks)
  Cost-effectiveness analysis of the FP-AF telerehabilitation program compared to conventional care assessed by data from EPR and databases at Region Midt & Viborg, Skive and Silkeborg Municipalities.
Cost-effectiveness analysis of the FP-AF telerehabilitation program compared to conventional care | Both intervention and control group: At the end of telerehabilitation (16 weeks) and at end follow up (28 weeks)
  Measured by European Quality og life - 5 Dimensions (EQ-5D) questionnaire. The questionaire is used to assess HRQoL and is comprised of 5 questions ranging from 1-5, with a lower score indicating a better outcome, and a higher score indicating a worse outcome. The questionnaire also has a question ranging from 0-100, with a lower score indicating a worse outcome and a higher score indicating a better outcome. The maximum score a patient can achieve in the questionnaire is 1, which indicates the best health state.
Patterns in multiparametric clinical monitoring | Intervention group: At the end of telerehabilitation (16 weeks).
  Data from devices for measuring blood pressure (mmHG) (systolic and diastolic) to analyze and identify correlations in multiparametric data.
Patterns in multiparametric clinical monitoring | Intervention group: At the end of telerehabilitation (16 weeks).
  Data from devices for measuring steps to analyze and identify correlations in multiparametric data.
Patterns in multiparametric clinical monitoring | Intervention group: At the end of telerehabilitation (16 weeks).
  Data from devices for measuring Electrocardiogram (ECG) to analyze and identify correlations in multiparametric data.
Patterns in multiparametric clinical monitoring | Intervention group: At the end of telerehabilitation (16 weeks).
  Data from devices for measuring weight (kilograms) to analyze and identify correlations in multiparametric data.
Patterns in multiparametric clinical monitoring | Intervention group: At the end of telerehabilitation (16 weeks).
  Data from devices for measuring pulse (numbers per minute) to analyze and identify correlations in multiparametric data.
Patterns in multiparametric clinical monitoring | Intervention group: At the end of telerehabilitation (16 weeks).
  Data from devices for measuring sleep (numbers of hours per night) to analyze and identify correlations in multiparametric data.
Future governance and infrastructure for telerehabilitation of AF patients | Intervention group: At the end of telerehabilitation (16 weeks)
  Interviews with patients and stakeholders

CONTACTS AND LOCATIONS:
Overall Officials: Birthe Dinesen, MSc, Ph.D, Principal Investigator — Aalborg University; Dorthe Svenstrup, MD, Ph.D, Study Director — Central Jutland Regional Hospital, Viborg; Lars Frost, MD, Ph.D, DMSc, Study Director — Central Jutland Regional Hospital, Silkeborg
Locations (1):
- Central Jutland Regional Hospital, Viborg and Silkeborg, Denmark

IPD SHARING:
Plan to Share IPD: No
No plan for sharing protocol as we are applying for patent.

REFERENCES:
- [Derived] Dinesen B, Albertsen AE, Joensen EDR, Spindler H, Jensen KM, Kidholm K, Frost L, Dittman L, Gunasegaram M, Johnsen SP, Jochumsen MR, Svenstrup D. Future Patient-Telerehabilitation of Patients With Atrial Fibrillation: Protocol for a Multicenter, Mixed Methods, Randomized Controlled Trial. JMIR Res Protoc. 2025 Feb 18;14:e64259. doi: 10.2196/64259. PMID 39965197
- See also: Read more about the trial at the homepage for the Laboratory for Welfare Technology - Digital health & rehabilitation, Aalborg University — https://www.labwelfaretech.com/fp/af/